CLINICAL TRIAL: NCT04462068
Title: ACE and HLA Genotypes Predict Severity and Disease Progression in Danish Sarcoid Patients
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: SAR3
Record Dates: First submitted 2020-05-11; First posted 2020-07-08 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-05

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sarcoidosis is a multisystem granulomatous disease of unknown cause histologically characterized by noncaseating granulomas. Genetic factors affect disease course, which is highly variable and difficult to predict.

This study aims to evaluate the predictive value of ACE and HLA genotypes on disease severity and progression in Danish patients with sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoidosis
* Signed informed consent

Exclusion Criteria:

* Inability or unwillingness to adhere to the study
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sarcoidosis seen in Department of Respiratory Diseases, Aarhus Denmark
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Time to initiation of treatment | 1 year from diagnosis
  Time to initiation of systemic immunosuppression for sarcoidosis

SECONDARY OUTCOMES:
Number of participants with extrapulmonary organ involvement | 1 year from diagnosis
  Number of participants diagnosed with extrapulmonary organ involvement
Change in FEV1 | 1 year
  Increase/ decline/ no change in FEV1
Change in FVC | 1 year
  Increase/ decline/ no change in FVC
Change in diffusion capacity | 1 year
  Increase/ decline/ no change in diffusion capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital. Dep. of Respiatory Diseases and Allergology, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided